CLINICAL TRIAL: NCT05941741
Title: Induction Chemotherapy Combined With Low-dose Radiation Plus Cadonilimab in Loco-regionally Advanced Nasopharyngeal Carcinoma: a Multi-center, Open-label, Randomized Controlled Phase III Clinical Trial
Brief Title: IC Plus Low-dose Radiation Plus Cadonilimab in LANPC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low-dose RT in NPC
Record Dates: First submitted 2023-07-01; First posted 2023-07-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma; Immune Checkpoint Inhibitor; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy; Induction Chemotherapy; Gemcitabine; Cisplatin; Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose RT plus ICI (Experimental): Patients will receive induction chemotherapy plus low-dose radiotherapy and immuce checkpoint inhibitor then followed by concurrent chemoradiotehrapy.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Chemotherapy; Biological: Immune checkpoint inhibitor; Radiation: Low-dose radiotherapy
- IC+CCRT (Active Comparator): Patients will receive induction chemotherapy plus concurrent chemoradiotehrapy.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — All target volumes will be outlined slice by slice on the axial contrast-enhanced CT with MR fusion images in the treatment planning system. The target volumes are defined in accordance with the International Commission on Radiation Units and Measurements Reports 83. The prescribed dose is 70-72 Gy to PTVp (Planning target volume of the primary tumor), 64-70 Gy to PTVn (Planning target volume of the lymph node), 60- 64Gy to PTV1 (High-risk planning target volume), and 54-58 Gy to PTV2 (Low-risk planning target volume) in 30-32 fractions.
  Other Names: IMRT
Drug: Chemotherapy — Induction chemotherapy: gemcitabine and cisplatin, Q3W, 3 cycles Concurrent chemotherapy: cisplatin, Q3W, 2-3 cycles
  Other Names: Induction chemotherapy; Concurrent chemotherapy; Gemcitabine; Cisplatin
Biological: Immune checkpoint inhibitor — Cadonilimab: 10mg/kg, Q3W, 3 cycles
  Other Names: Cadonilimab; AK104; PD-1/CTLA-4 inhibitor
  Arms: Low-dose RT plus ICI
Radiation: Low-dose radiotherapy — Low-dose radiotherapy will be performed to study group, with the use of IMRT.
  Arms: Low-dose RT plus ICI

SUMMARY:
This is a multi-center, open-label, randomized controlled phase III clinical trial in primary diagnosed loco-regionally advanced nasopharyngeal carcinoma (NPC) patients. The purpose of this study is to evaluate the efficacy of induction chemotherapy (IC) combined with low-dose radiation and immune checkpoint inhibitor (ICI) followed by concurrent chemoradiotherapy (CCRT) versus IC+CCRT, and compare the treatment-related adverse events and quality of life in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal non-keratinizing carcinoma (WHO II/III);
* All genders, range from 18-70 years old;
* ECOG score 0-1;
* Clinical stage T4N1M0 and T1-4N2-3M0 (AJCC/UICC 8th);
* Not received radiotherapy, chemotherapy and other anti-tumor treatment (including immunotherapy);
* No contraindications to chemotherapy, radiotherapy or immunotherapy;
* Adequate organ function: white blood cell count ≥ 4×109/L, neutrophile granulocyte count ≥ 1.5×109/L, hemoglobin ≥ 9g/L, platelet count ≥ 100×109/L; alanine aminotransferase or aspartate aminotransferase < 2.5×upper limit of normal; blood urea nitrogen or creatinine ≤ 1.5×upper limit of normal or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Sign the consent form.

Exclusion Criteria:

* Distant metastases;
* Keratinized squamous cell carcinoma or basal cell like squamous cell carcinoma;
* Have or are suffering from other malignant tumors;
* Participating in other clinical trials;
* Pregnancy or lactation;
* Have uncontrolled cardiovascular disease;
* Severe complication, eg, uncontrolled hypertension;
* Mental disorder;
* Drug or alcohol addition;
* Do not have full capacity for civil acts.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 years
  From the date of randomization to local or regional recurrence, distant metastasis or any death

SECONDARY OUTCOMES:
Overall survival | 3 years
  From the date of randomization to any death, with patients unavailable for follow-up censored at the date of last follow-up
Local recurrence-free survival | 3 years
  From the date of randomization to local recurrence or any death
Regional recurrence-free survival | 3 years
  From the date of randomization to regional recurrence or any death
Distant metastasis-free survival | 3 years
  From the date of randomization to distant metastasis or any death
Acute toxicities | From the start of treatment until 3 months post treatment
  Assessed with CTCAE v5.0
Late toxicities | 3 years post treatment
  Assessed with RTOG/EORTC
Quality of life score | Through study completion, an average of 3 years
  Assessed with EORTC-Quality of life questionnaire-C30 version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn